CLINICAL TRIAL: NCT00318071
Title: A Multinational Controlled Registry to Evaluate the Concentric Merci Retriever System (Mechanical Embolus Removal in Cerebral Ischemia [MERCI™])
Brief Title: Multi MERCI (Mechanical Embolus Removal in Cerebral Ischemia [MERCI™])
Acronym: Multi-MERCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stryker Neurovascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INT-LR-001
Record Dates: First submitted 2005-07-14; First posted 2006-04-26 (Estimated); Last update posted 2014-11-07 (Estimated); Status verified 2014-11

CONDITIONS: Ischemic Stroke
Keywords: Stroke; Ischemic; Thrombus; Embolectomy; Thrombectomy; Merci; Concentric; Embolus; Embolism; Mechanical
MeSH Terms: conditions — Ischemic Stroke; Stroke; Ischemia; Thrombosis; Embolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Treatment arm patients had at least one Merci Retriever deployed
  Interventions: Device: Merci Retriever

INTERVENTIONS:
Device: Merci Retriever — For patients eligible to participate in the trial, the operating physician initiated treatment with the Merci L5 Retriever to remove large vessel thrombotic occlusion and recanalization of the vessel. Subsequent treatment could be made with Merci X6 or X5 Merci Retrievers.
  Large vessel arteries are defined as internal carotid, middle cerebral M1/M2 segments, basilar, and vertebral arteries.
  Recanalization was defined as TIMI II or TIMI III per angiography.

SUMMARY:
The primary objectives of the Multi MERCI trial were:

* to evaluate the addition of the Merci L5 Retriever
* additionally permit use of the Merci Retrieval System in the setting of persistent clot following IV t-PA treatment (use in the 0-8 hour window for patients ineligible for IV t-PA was also permitted)

DETAILED DESCRIPTION:
Per the Multi MERCI protocol, up to 230 patients could be treated at up to 30 centers.

The intended trial indication for the Merci L5 Retriever was to restore blood flow in the neurovasculature by removing thrombus in patients experiencing ischemic stroke. Patients that were contraindicated or failed treatment with intravenous t-PA were allowed to be enrolled under the Multi MERCI protocol.

Per the Multi MERCI protocol, following inclusion of the Merci L5 Retriever the operating physician was required to initiate treatment with the Merci L5 Retriever. At the physician's discretion, subsequent passes could be made with the Merci L5 Retriever, Merci X6 Retriever and/or Merci X5 Retriever.

Adverse events were adjudicated by an independent Data Safety and Monitoring Board (Capital DSMB).

ELIGIBILITY:
Inclusion Criteria:

* Angiographically confirmed large vessel ischemic stroke (occlusion may include the following: internal carotid artery (ICA), M1/M2, vertebral, or basilar arteries)
* Intervention is able to be performed within 8 hours of symptom onset
* Patients > 18 years of age
* NIHSS score 8+
* Failed IV t-PA treatment or contraindicated for IV t-PA

Exclusion Criteria:

* International Normalized Ratio (INR) > 3.0
* Platelet count < 30,000
* Heparin use in previous 24 hours with PTT > 2X normal
* Baseline bloog glucose < 50 mg/dL
* Baseline computed tomography (CT) showing mass effect with midline shift
* Severe sustained hypertension (SBP > 185 or DBP > 110) that cannot be controlled with medication
* Patient is pregnant, has anticipated life expectancy < 3 months, or has severe allergy to contrast medium
* Arterial stenosis > 50% proximal to embolus
* Excessive arterial tortuosity that precludes the study device from reaching the target area

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2004-01; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Revascularization success; Rates of device-related serious adverse events | post-procedure

SECONDARY OUTCOMES:
modified Rankin scores | 90-day
mortality | 90-day
Symptomatic hemorrhage rate | 24 hour post procedure

CONTACTS AND LOCATIONS:
Overall Officials: Wade S Smith, MD, PhD, Principal Investigator — University of California, San Francisco

REFERENCES:
- [Result] Smith WS, Sung G, Saver J, Budzik R, Duckwiler G, Liebeskind DS, Lutsep HL, Rymer MM, Higashida RT, Starkman S, Gobin YP; Multi MERCI Investigators; Frei D, Grobelny T, Hellinger F, Huddle D, Kidwell C, Koroshetz W, Marks M, Nesbit G, Silverman IE. Mechanical thrombectomy for acute ischemic stroke: final results of the Multi MERCI trial. Stroke. 2008 Apr;39(4):1205-12. doi: 10.1161/STROKEAHA.107.497115. Epub 2008 Feb 28. PMID 18309168
- [Result] Smith WS. Safety of mechanical thrombectomy and intravenous tissue plasminogen activator in acute ischemic stroke. Results of the multi Mechanical Embolus Removal in Cerebral Ischemia (MERCI) trial, part I. AJNR Am J Neuroradiol. 2006 Jun-Jul;27(6):1177-82. PMID 16775259
- [Result] Flint AC, Duckwiler GR, Budzik RF, Liebeskind DS, Smith WS; MERCI and Multi MERCI Writing Committee. Mechanical thrombectomy of intracranial internal carotid occlusion: pooled results of the MERCI and Multi MERCI Part I trials. Stroke. 2007 Apr;38(4):1274-80. doi: 10.1161/01.STR.0000260187.33864.a7. Epub 2007 Mar 1. PMID 17332445
- [Result] Lutsep HL, Rymer MM, Nesbit GM. Vertebrobasilar revascularization rates and outcomes in the MERCI and multi-MERCI trials. J Stroke Cerebrovasc Dis. 2008 Mar-Apr;17(2):55-7. doi: 10.1016/j.jstrokecerebrovasdis.2007.11.003. PMID 18346645
- [Derived] Shi ZS, Liebeskind DS, Xiang B, Ge SG, Feng L, Albers GW, Budzik R, Devlin T, Gupta R, Jansen O, Jovin TG, Killer-Oberpfalzer M, Lutsep HL, Macho J, Nogueira RG, Rymer M, Smith WS, Wahlgren N, Duckwiler GR; Multi MERCI, TREVO, and TREVO 2 Investigators. Predictors of functional dependence despite successful revascularization in large-vessel occlusion strokes. Stroke. 2014 Jul;45(7):1977-84. doi: 10.1161/STROKEAHA.114.005603. Epub 2014 May 29. PMID 24876082
- [Derived] Liebeskind DS, Flint AC, Budzik RF, Xiang B, Smith WS, Duckwiler GR, Nogueira RG; MERCI and Multi-MERCI Investigators. Carotid I's, L's and T's: collaterals shape the outcome of intracranial carotid occlusion in acute ischemic stroke. J Neurointerv Surg. 2015 Jun;7(6):402-7. doi: 10.1136/neurintsurg-2014-011231. Epub 2014 May 1. PMID 24789707
- See also: Concentric Medical Website — http://www.concentric-medical.com